CLINICAL TRIAL: NCT01834105
Title: Study on the Molecular Mechanism of Postmenopausal Osteoporosis With Kidney Yin Deficiency Syndrome From CLCF1 Interventing on JAK-STAT Signaling Pathways
Brief Title: Molecular Mechanism of POP Kidney Yin Deficiency Syndrome From the Interventional Effects of CLCF1
Acronym: pop
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Academy of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 81173280
Record Dates: First submitted 2013-04-14; First posted 2013-04-17 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Postmenopausal osteoporosis; Kidney Yin deficiency syndrome; Liuwei dihuang pill; CLCF1; JAK - STAT signal pathway
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Crisponi syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liuwei Dihuang Pills (Experimental)
  Interventions: Drug: Liuwei Dihuang Pills

INTERVENTIONS:
Drug: Liuwei Dihuang Pills

SUMMARY:
This study use RT-PCR and Western Blot technique to detect the expression of CLCF1 mRNA and protein in POP Kidney Yin deficiency group and healthy group to verify the relevance between CLCF1 and POP the kidney Yin deficiency syndrome.Through siRNA and overexpression,observe the mRNA and protein 's expression of CBP、JAK1、STAT4 and the protein phosphorylation of JAK1、STAT4 in JAK-STAT signal to reveal the CLCF1 regulate the CBP's mechanism.Use the Liuwei Dihuang Pills to detect the effect of treatment ,compare use or not the Liuwei Dihuang Pills to detect the mRNA and protein 's expression of CLCF1、CBP etc.Aim to clarify the POP kidney Yin deficiency molecular mechanism.

ELIGIBILITY:
Inclusion Criteria:

* The Participants who volunteer to be test subjects, and can accept experimental drugs, and promise to finish the course should sign the informed consent.
* Female ages 45 to 75 had gone through natural menopause before two years
* In accordance with the western medicine diagnostic criteria of osteoporosis and belong to kidney Yin deficiency syndrome differentiation of traditional Chinese medicine certificate;
* In accordance with the western medicine diagnostic criteria;
* In accordance with TCM diagnostic methods; .If any of the above answers are no, The subjects couldn't in the study.

Exclusion Criteria:

* Do not accord with standard of the western medicine diagnosis and TCM diagnostic methods
* Age: <44 and > 76 years old;
* With hyperparathyroidism, osteomalacia, rheumatoid arthritis, multiple myeloma and other serious complications such as secondary osteoporosis; Late or deformity, disability, loss of labor;
* With cardiovascular, cerebrovascular, liver, kidney and hematopoietic system and other serious primary diseases;
* Psychosis or alzheimer's patients;
* Nearly three months, the use of hormone replacement therapy (HRT) and taking calcitonin, nearly six months has used double phosphonic acid salt for 15 days, etc.;
* This medicine allergic constitution or composition of known to have allergies;
* In a critical condition, It's difficult to make exact evaluators to efficacy and safety of the new drugs;

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
osteoporosis treatment within six months of study enrollment | Liuwei Dihuang Pills therapy (up to six months)

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Institute of Trational Chiness Medicine, Fuzhou, Fujian, China